CLINICAL TRIAL: NCT05949437
Title: The Effect of Yoga Breathing Exercises Versus Aerobic Exercise on Hematological Parameters in Iron Deficiency Anemic Females
Brief Title: Effect of Yoga Breathing Exercises Versus Aerobic Exercise on Hematological Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shokry Mahmoud Youssef Mohamed (Other)
Responsible Party: Sponsor-Investigator, Shokry Mahmoud Youssef Mohamed, Assistant lecturer of physical therapy for Internal Medicine and Geriatrics, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004556
Record Dates: First submitted 2023-06-27; First posted 2023-07-18 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-07

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (I) (Experimental): consists of 30 patients with iron deficiency anemia and will receive medical treatment of anemia, Dietary advices and 50 minutes yoga therapy 6 days a week for 12 weeks
  Interventions: Other: Yuga
- Group (II) (Other): consists of 30 patients with iron deficiency anemia and will receive medical treatment for anemia, Diet advices and 30 minutes of aerobic exercises in form of treadmill according to the target exercise heart rate for 12 weeks.
  Interventions: Other: Aerobic exercises

INTERVENTIONS:
Other: Yuga — Traditional yoga body posture for 15 minutes, yoga breathing exercises for 30 minutes and meditation for 5 minutes for 12 weeks
  Arms: Group (I)
Other: Aerobic exercises — in form of treadmill according to the target exercise heart rate for 12 weeks
  Arms: Group (II)

SUMMARY:
Is there effect of yoga breathing exercises versus aerobic exercise on hematological parameters in iron deficiency anemic females?

The purpose of the study is to investigate the effect of yoga breathing exercises versus aerobic exercise on hematological parameters in iron deficiency anemic females

DETAILED DESCRIPTION:
60 patients with iron deficiency anemia and will receive medical treatment of anemia and Dietary advice for 12 weeks . thirty patient from the 60 patients will receive yoga therapy and 50 minutes yoga therapy 6 days a week for 12 weeks while the other 30 patients will receive aerobic exercise for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Sixty female patients referred with iron deficiency anemia
2. Their age will be ranged from 30-40 years old.
3. All patients have a history of anemia.
4. All patients should be medically stable.
5. The body mass index (BMI) ranged from 25:29.9 Kg/m2
6. Number of parity not exceed 3 times.
7. Period of menses from 3-5 days

Exclusion Criteria:

1. Patients with cognitive impairments.
2. All types of anemia except iron deficiency anemia
3. patients with hearing problems.
4. patients with Diabetes, Hypertension.
5. Patients with Musculoskeletal, Neurological, Cardiovascular and Respiratory problems
6. patients with mental problems.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
serum iron level | it will be measured after 12 weeks
  it will be measured in serum from complete blood picture. Reference range from 50 till 212 ug/dl. Number of participants are 60 females.
ferritin level | it will be measured after 12 weeks
  it will be measured in serum from iron profile. Reference range from 10 till 158 ng/ml. Number of participants are 60 females.
iron binding capacity level | it will be measured after 12 weeks
  it will be measured in serum from iron profile. Reference range from 250 till 400 ug/dl. Number of participants are 60 females.
count of red blood cells | it will be measured after 12 weeks
  it will be measured in serum from complete blood picture. Reference range from 3.80 till 4.80 million cell/cmm. Number of participants are 60 females.
Hemoglobin level | it will be measured after 12 weeks
  it will be measured in serum from complete blood . picture. Reference range from 12 till 15 g/dl. Number of participants are 60 females.
hematocrite level | it will be measured after 12 weeks
  it will be measured in serum from complete blood picture. Reference range from 36% till 45%. Number of participants are 60 females.
lymphocytes level | it will be measured after 12 weeks
  it will be measured in serum from differential white cell count. Reference range absolute from 1000 till 4000 and relative from 20% till 45%. Number of participants are 60 females.

SECONDARY OUTCOMES:
six minute walking distance | it will be measured after 12 weeks
  The six minute walking distance is measured using six Minute Walk Test which is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  The tools are used include 30 meters corridor,2 cones,stopwatch,chair,mechanical lap counter and sphygmomanometer Number of participants are 60 females.
The fatigue severity scale(FSS) | it will be measured after 12 weeks
  The FSS questionnaire contains nine statements that rate the severity of your fatigue symptoms. Read each statement and circle a number from 1 to 7, based on how accurately it reflects your condition during the past week and the extent to which you agree or disagree that the statement applies to you.
  A total score of less than 36 suggests that you may not be suffering from fatigue.
  A total score of 36 or more suggests that you may need further evaluation by a physician.
  Number of participants are 60 females.

CONTACTS AND LOCATIONS:
Overall Officials: shoukry MA youssef, ass lecturer, Principal Investigator — 6 october University
Locations (1):
- October 6 university, Giza, Egypt